CLINICAL TRIAL: NCT04856150
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of Q-1802 in Patients With Advanced Solid Tumors
Brief Title: A Study of Q-1802 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: QureBio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Qure-1802-101
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Q-1802 (Experimental): Q-1802 dose exploration and Q-1802 dose extension
  Interventions: Drug: Q-1802

INTERVENTIONS:
Drug: Q-1802 — Q-1802 will be administered intravenously.

SUMMARY:
Q-1802 is a bispecific antibody targeting both the tumor-specific antigen Claudin 18.2 and the immune checkpoint PD-L1. This is a multi-center, single-arm, open-label design to evaluate the safety and tolerance of Q-1802 in patients with advanced solid tumors, together with an assessment of pharmacokinetic characteristics and efficacy. The study consisted of two compartments: the dose-exploration stage and the dose-extension stage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥18 years and ≤75 years.
* Patients with at least one measurable lesion per RECIST (v1.1) (applicable to the dose-extension stage).
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1 at screening and no deterioration occurs within two weeks before enrollment.
* Life expectancy period ≥ 12 weeks.
* Patients who have sufficient baseline organ function and whose laboratory data meet the following criteria (receiving no treatment of blood transfusions, albumin, recombinant human thrombopoietin, or colony-stimulating factor within 14 days before the first dose of this study).
* Patients with advanced gastric mucinous adenocarcinoma, advanced ovarian mucinous carcinoma or other dominant tumors participating in the dose-extension stage must provide eligible tumor tissue samples for biomarker detection; if subjects agree, tumor tissue samples should also be provided during the dose-exploration stage.

Exclusion Criteria:

* Patients who have received any prior PD-1/PD-L1 antibody therapy (applicable to the dose-exploration stage).
* Patients with uncontrolled blood pressure (systolic blood pressure ≥ 150 mm Hg and/or diastolic blood pressure ≥ 100 mm Hg) or previous hypertensive crisis or hypertensive encephalopathy.
* Patients with active peptic ulcer, gastric outlet obstruction or persistent recurrent vomiting.
* Patients with a history of monoclonal antibody allergic reaction.
* Patients who are considered ineligible by the investigator due to any other severe, acute or chronic disease or other causes that the investigator considers could affect the patient's participation or assessment in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | 28 days
  Incidence of dose limiting toxicities(DLTs). A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle with Q-1802.

SECONDARY OUTCOMES:
Plasma concentration (Cmax) | 70 days
  Highest observed plasma concentration of Q-1802
Time to achieve Cmax (Tmax) | 70 days
  Time of highest observed plasma concentration of Q-1802
Area under the plasma concentration-time curve (AUC) | 70 days
  Area under the plasma concentration time curve of Q-1802
PD-L1 receptor occupancy rate (RO) | 70 days
  PD-L1 receptor occupancy rate (RO) on the surface of T lymphocytes in peripheral blood at different time points of Q-1802
Number of participants with treatment-related adverse events(TRAE) | 70 days
  TRAE is defined as the AEs that the casual relationship of the AE is ralated to Q-1802.
Objective response rate (ORR) | 70 days
  ORR is defined as proportion of participants with complete response, partial response (CR+PR).
Progression-free survival (PFS) | 70 days
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first.
Duration of response ( DCR ) | 70 days
  DCR is defined as proportion of participants with complete response, partial response, stable disease (CR+PR+SD).
Duration of response ( DOR ) | 70 days
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing cancer hospical, Beijing
  - West China Second University Hospical, Sichuan University, Chengdu
  - Fudan University Shanghai Cancer Center, Shanghai
  - PKUCare Luzhong Hospital, Zibo